CLINICAL TRIAL: NCT02351947
Title: Structural and Functional Brain Changes in Response to Post-Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louis Stokes VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Svetlana Pundik, M.D., Director, Brain Plasticity and Neurorecovery Laboratory, Louis Stokes VA Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B6636W
Record Dates: First submitted 2014-12-16; First posted 2015-01-30 (Estimated); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Cerebrovascular Accident
Keywords: stroke; Cerebrovascular accident; rehabilitation; motor learning; fMRI; plasticity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- persons with chronic stroke (Experimental): upper limb rehabilitation for chronic stroke
  Interventions: Other: upper limb rehabilitation for chronic stroke
- Healthy, age matched control group (No Intervention): Healthy aged match control group undergoing MRI/EEG testing

INTERVENTIONS:
Other: upper limb rehabilitation for chronic stroke — subjects in this group will receive upper limb motor learning rehabilitation and undergo fMRI/EEG testing as well as testing of motor function (AMAT and FM).
  Arms: persons with chronic stroke

SUMMARY:
The purpose of this research study is to improve methods for evaluation of brain changes during motor learning for patients with stroke, who have difficulty performing daily tasks with their arm and hand. The methods for evaluation of brain changes will consist of the combination of magnetic resonance imaging (MRI) and electroencephalography (EEG).

DETAILED DESCRIPTION:
A third of American Veterans is left with moderate to severe motor deficits after stroke. Intensive rehabilitation can resolve some of these deficits. Motor function restoration is associated with and dependent on reorganization of neuronal networks (i.e. plasticity). However, our understanding of human brain plasticity during functional recovery is incomplete. Furthermore, it is unknown what patterns of structural brain changes are associated with greater gains in motor function as a result of motor learning therapy. The main objective of the study is to characterize the reorganization of brain structure and function that is associated with greater gains in motor function following restorative rehabilitation for chronic survivors. This will further our understanding of recovery after brain injury and subsequently assist in more accurately directing rehabilitation therapies to produce the best possible outcomes.

The two hypotheses are: I. There is reorganization of both movement control brain regions and pathways between regions that is associated with functional motor recovery in response to intensive motor learning after stroke; and II. For stroke victims with upper extremity deficits, motor recovery is associated with changes in the sequential timing of activity across cortical regions.

Design and Methods. A cohort of chronic stroke survivors with upper extremity deficits will be treated by our intensive multimodal 12-week motor learning program. Brain imaging (functional Magnetic Resonance Imaging (fMRI) and Diffusion Tensor Imaging (DTI)) and neurophysiological (Electroencephalogram (EEG)) studies as well as functional motor tests (Arm Motor Activity test and Fugl-Meyer Coordination test) will be obtained before and after the treatment. Age-matched control subjects will be evaluated as well. DTI/fMRI and EEG/fMRI combination techniques will be used to determine changes in brain structure and function as a result of the treatments. A regression analysis will determine which brain structure parameters can predictor greater motor function gains.

ELIGIBILITY:
Inclusion Criteria for chronic stroke patients:

1. Medically stable and at least 6 months post ischemic stroke.
2. Inability to use upper limb for functional tasks
3. Sufficient endurance to participate in rehabilitation
4. Cognition sufficiently intact to give valid informed consent to participate
5. Ability to follow two stage commands
6. Trace or better contraction of the following muscles: finger flexors, wrist flexors and extensors, shoulder flexors or abductors, shoulder horizontal abductors, scapular retractors
7. Muscle tone of fingers, wrist and elbow flexors ≤3 (Ashworth scale)
8. Age > 21

Exclusion Criteria

1. Acute or progressive cardiac, renal, respiratory, neurological disorders or malignancy
2. Active psychiatric diagnosis or psychological condition
3. Lower motor neuron damage or radiculopathy
4. Hand grasp and release sufficient to grasp 4 oz. can, lift 12 inches, replace it in original position and release grasp within 1-2 seconds of the time of the unaffected extremity
5. Absent position sense at elbow or wrist
6. More than one ischemic strokes or stroke affecting both sides
7. Metal implants, pacemaker, claustrophobia, or inability to operate the MRI patient call button

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
functional MRI during movement of the shoulder and elbow | up to 3 months
  MRI allows for observation of the internal structures of the body using a magnetic field and radiowaves. We will measure activation voxel count in response to training.
Electroencephalography (EEG) during movement of the shoulder and elbow | Day 1 and following 3 months of intervention
  EEG is used to record electrical signals released by the brain. We will assess changes in the movement related cortical potentional (MRCP, measured in microvolts) in response to training.

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana Pundik, M.D., Principal Investigator — Louis Stokes VA Medical Center
Locations (1):
- Louis Stokes Cleveland Department of Veterans Affairs Medical Center, Cleveland, Ohio, United States